CLINICAL TRIAL: NCT01669538
Title: Repurposing Cholinesterase Inhibitors for Smoking Cessation.
Brief Title: Effect of Galantamine on Short-term Abstinence
Acronym: GAL-K
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); National Center for Research Resources (NCRR) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 815789; UPCC15912 (Other: Abramson Cancer Center of the University of Pennsylvania); K23DA035295 (NIH); NCT01845961 (obsolete NCT alias)
Record Dates: First submitted 2012-08-16; First posted 2012-08-21 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Tobacco Use Disorder
Keywords: Galantamine; Nicotine Bitartrate; Nicotine Tartrate; Nicotine dependence; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Galantamine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Galantamine (Experimental): Galantamine hydrobromide-ER (extended release) is currently marketed for the treatment of Alzheimer's disease. The dosing regimen follows the FDA-approved guidelines. For the first week of study treatment, participants will take 8mg daily of galantamine-ER, preferably with food. 8mg is the lowest dose and this period is designed to introduce the medication into their system. After the initial week, participants will increase their daily dose to 16mg. They will remain on 16mg daily until the end of the treatment period for a total of 23 days on active study medication.
  Galantamine will be purchased, encapsulated, and packaged into blister packs by the Investigational Drug Service at the University of Pennsylvania. Both active medication and placebo will look identical.
  Interventions: Drug: Galantamine
- Placebo (Placebo Comparator): Participants assigned to the placebo (sugar pill) arm will take one capsule daily, preferably with food, for a total of 23 days. They will follow the same instructions and complete the same procedures as those in the active treatment.
  Placebo ingredients (sucrose filler and gel capsules) will be purchased, encapsulated, and packaged into blister packs by the Investigational Drug Service at the University of Pennsylvania. Both active medication and placebo will look identical.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galantamine
  Other Names: Galantamine hydrobromide ER; Razadyne ER
  Arms: Galantamine
Drug: Placebo
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled study to test whether a medication called galantamine (Brand Name: Razadyne) will help smokers quit and whether it reduces cognitive problems that smokers experience during a quit attempt.

DETAILED DESCRIPTION:
Galantamine, an FDA-approved treatment for Alzheimer's disease, is used to treat cognitive impairment by enhancing acetylcholine through inhibition of the enzyme, acetylcholinesterase. We propose randomized double-blind placebo-controlled study of short-term (23 days) treatment with galantamine.

Eighty chronic smokers will complete a validated procedure for screening new medications. An equal number of subjects will be assigned to one of two groups: galantamine-ER or placebo. Participants in both groups will take one capsule each day and follow the same procedures. This is not a cross-over trial.

For participants in the galantamine group, following an initial 1-week drug run-up phase (8mg daily of galantamine-ER), the medication dose will be increased to 16mg daily of galantamine-ER for the remainder of the study (up to Day 23).

On Day 15, smokers will begin a mandatory 24-hour abstinence period, which will be followed by a programmed smoking lapse on Day 16. Smokers will then be instructed to abstain for the following 7 days (observed abstinence). Following completion of the study, participants will be offered standard smoking cessation treatment.

On Days 0 (Baseline), 14, and 16, subjects will perform the following computer tasks: a working memory task (Visual/Spatial N-Back), sustained attention tasks (Penn Continuous Performance Task [PCPT-nl] and XO Reaction Time Task), a recall memory task (Word Recognition), an interference control task (Stroop test), and a response inhibition task (Stop Signal Task).

The primary outcome is to identify changes in behavioral performance and subjective symptoms following two weeks treatment of galantamine and after 24 hours of abstinence, compared to baseline.

This study will provide information about the role of the cholinergic system during brief abstinence and whether enhancing acetylcholine reduces abstinence-induced cognitive symptoms that promote smoking relapse. Information obtained in this study may further establish cognitive performance measures as endophenotypes for nicotine dependence.

ELIGIBILITY:
Inclusion Criteria:

1. Smokers who are between 18 and 60 years of age who self-report smoking at least 10 cigarettes (menthol and non-menthol) per day for at least the last 6 months.
2. Interest in quitting smoking in the next 2 to 6 months.
3. Healthy as determined by the Study Physician, based on a medical evaluation including medical history and physical examination, and psychiatric evaluation.
4. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form.
5. Women of childbearing potential must consent to use a medically accepted method of birth control while participating in the study (e.g., condoms and spermicide, oral contraceptive, Depo-provera injection, contraceptive patch, tubal ligation).

Exclusion Criteria:

1. Smoking behavior

   1. Use of chewing tobacco, snuff, and/or snus.
   2. Current enrollment in a smoking cessation program, or use of other smoking cessation medications in the last month or plans to do either in the next 2 months.
   3. Provide a carbon monoxide (CO) breath sample reading less than 10 parts per million (ppm) at either the Intake or Baseline visits.
2. Alcohol/Drugs

   1. Lifetime history of substance abuse (other than nicotine) and/or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, stimulants, PCP, benzodiazepines, or study-prohibited medications/recreational drugs) as determined by self-report during the phone screen and/or through the MINI during the Intake visit.
   2. Current alcohol consumption that exceeds 25 standard drinks/week over the past 6 months.
   3. Providing a breath alcohol concentration (BrAC) reading of greater than or equal to 0.01 at the Intake, Baseline, or Testing Days.
   4. A positive urine drug screen for cocaine, amphetamines, methamphetamines, benzodiazepines, PCP, methadone, barbiturates, and opiates at the Intake visit, Baseline visit, or the Testing days.
3. Medical

   1. Women who are pregnant, planning a pregnancy in the next 3 months, or lactating; all female subjects shall undergo a urine pregnancy test at the Intake visit and must agree in writing to use an approved method of contraception. Following enrollment, pregnancy tests will be conducted at the Baseline visit and Testing days for all female subjects of child-bearing potential.
   2. Diagnosis of Alzheimer's Disease or dementia.
   3. Current treatment of cancer or diagnosed with cancer (except basal cell carcinoma) in the past 6 months.
   4. Liver/kidney failure, peptic ulcer disease, benign prostate hypertrophy.
   5. Asthma or chronic obstructive pulmonary disease (COPD).
   6. History (last 6 months) of abnormal heart rhythms, tachycardia and/or cardiovascular disease (stroke, angina, heart attack). These conditions will be evaluated on a case by case basis by the Study Physician/Health Care Provider.
   7. Serious or unstable disease within the past 6 months, as determined by the Study Physician/Health Care Provider.
   8. Clinically significant abnormalities within physical examination and vital signs at Medical Screen. Abnormalities will be assessed by the Study Physician/Health Care Provider and eligibility will be determined on a case-by-case basis.
   9. Any impairment (physical and/or neurological) including visual or other impairment preventing cognitive task performance.
   10. Uncontrolled high blood pressure (Systolic BP greater than 160 and/or Diastolic BP greater than 100).
   11. Hearing impairment, significant hearing loss (more than 20% in either ear), cochlear implants, or bi-lateral hearing aids.
   12. History of brain injury.
   13. History of epilepsy or a seizure disorder.
   14. Color Blindness.
   15. Low or borderline intellectual functioning - determined by receiving a score of less than 90 on the Shipley Institute of Living Scale (SILS) which correlates with the Wechsler Adult Intelligence Scale-Revised (WAIS-R) Estimated IQ Test (administered at the Intake visit).
4. Psychiatric Exclusions (determined by self-report on phone screen and/or through the MINI during the Intake visit)

   1. Current diagnosis of major depression. Persons with a history of major depression, in remission for 6 months or longer, are eligible, provided they are not excluded based on medications (below).
   2. Suicide risk score on MINI greater than 0.
   3. History or current diagnosis of schizophrenia, psychosis, and/or bipolar disorder.
   4. Current or past hypomanic/manic episode.
   5. Current or history of a diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD).
5. Medication

   1. Current use, recent discontinuation (within the last month) of any form of smoking cessation medications (i.e., Zyban, Wellbutrin, Wellbutrin SR, Chantix, nicotine replacement therapy).
   2. Current use or recent discontinuation (within the last 60 days) of any of the following:

      * Anti-anxiety or panic disorder medications.
      * Anti-psychotic medications.
      * Mood-stabilizers (e.g., Lithium, Lamictal/lamotrigine, Neurontin/gabapentin, Topamax/topiramate, valproic acid, Tegretol/carbamazepine).
      * Anti-depressants (e.g., Wellbutrin, MAOIs, SSRIs, tricyclic antidepressants).
      * Prescription stimulants (e.g., Provigil, Ritalin, Adderall).
      * Systemic Steroids (e.g., Prednisone).
      * Alzheimer's disease medications (e.g., Acetylcholinesterase inhibitors (ACIs), Aricept/donepezil, Exelon/rivastigmine, Tacrine, or memantine).
      * Parkinson's disease medications(e.g., Cogentin/benztropine).
      * Irritable bowel syndrome medication (e.g., Dicylomine/Bentyl).
      * Heart medications (e.g., quinidine or Procardia/nifedipine).
      * Peptic ulcer disease medication (e.g, Zantac/ranitidine).
      * Muscle relaxants (e.g., Soma/carisoprodol, Anectine/succinylcholine).
      * Anti-fungal medication (e.g., Nizoral/ketoconazole).
      * Anti-seizure medications (e.g., Ativan, Banzel, Carbatrol, Dilantin, Lamictal, Gabitril, Lyrica, Neurontin, Tegretol, Topamax).
      * COPD medication (e.g., Atrovent/Ipratropium Bromide).
      * Urinary retention medications (e.g., Duvoid/bethanechol, Proscar/finasteride, Avodart/dutasteride, Dibenzyline/phenoxybenzamine, Regitine/phentolamine).
      * Eye medication (e.g., Atropine).
   3. Daily use of any of the following:

      * Opiate-containing medications for chronic pain (Duragesic/fentanyl patches, Percocet, Oxycontin).
      * Medication for asthma (albuterol, Serevent, Combivent, Advair, Flovent, Azmacort, Symbicort).
   4. Known drug allergy to the study medication.

   Subjects will be instructed to refrain from using any study prohibited drugs/medications (both recreational and prescription) throughout their participation in the study. After final eligibility is confirmed, subjects who report taking contraindicated medication(s) over the course of the study period may only remain eligible if the Study Physician and/or Principal Investigator determines that the contraindicated medication(s) do/did not impact the study design, data quality, and/or subject safety/welfare. Subjects are permitted to take necessary prescription medications not included within the exclusion list during the study.
6. General exclusions

   1. Current, anticipated, or pending enrollment in another research program over the next 2-3 months that could potentially affect subject safety and/or the study data/design as determined by the Principal Investigator and/or Study Physician.
   2. Not planning to live in the area for the next two months.
   3. Any medical condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.
   4. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator.
   5. Completion of neurocognitive assessments and/or use of study medication(s) at the CIRNA in the past 6-months that could influence performance on study tasks as determined by the Principal Investigator.
   6. Not able to effectively communicate in English (reading, writing, speaking).
   7. Missing 2 or more consecutive sessions, or 3 or more sessions during the medication period.
   8. Missing 2 or more consecutive doses during the medication period.
   9. Missing 3 or more doses throughout the medication period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2012-08; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Ashare, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Interdisciplinary Research on Nicotine Addiction, University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 98 subjects who enrolled in the study, 16 were deemed ineligible to participate and therefore not assigned to a treatment arm (i.e., did not Start the study). Thus, 82 subjects Started the study.
Groups:
- Galantamine: Galantamine hydrobromide-ER (extended release) is currently marketed for the treatment of Alzheimer's disease. The dosing regimen follows the FDA-approved guidelines. For the first week of study treatment, participants will take 8mg daily of galantamine-ER, preferably with food. 8mg is the lowest dose and this period is designed to introduce the medication into their system. After the initial week, participants will increase their daily dose to 16mg. They will remain on 16mg daily until the end of the treatment period for a total of 23 days on active study medication.
  Galantamine will be purchased, encapsulated, and packaged into blister packs by the Investigational Drug Service at the University of Pennsylvania. Both active medication and placebo will look identical.
  Galantamine
- Placebo: Participants assigned to the placebo (sugar pill) arm will take one capsule daily, preferably with food, for a total of 23 days. They will follow the same instructions and complete the same procedures as those in the active treatment.
  Placebo ingredients (sucrose filler and gel capsules) will be purchased, encapsulated, and packaged into blister packs by the Investigational Drug Service at the University of Pennsylvania. Both active medication and placebo will look identical.
  Placebo
Period: Overall Study
Arm/Group | Galantamine | Placebo
Started | 40 | 42
Completed | 28 | 33
Not Completed | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galantamine | Placebo | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (11.3) | 42.8 (10.9) | 42.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 22 | 29 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 38 | 40 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 26 | 50
  White | 13 | 9 | 22
  More than one race | 2 | 5 | 7
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 42 | 82
Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Self-report measure of nicotine dependence on a scale from 0 to 10 with 0 being not at all dependent and 10 being highly dependent.
  units on a scale | 5.1 (1.5) | 5.4 (1.8) | 5.2 (1.7)
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes] | 15.2 (4.7) | 15.5 (6.9) | 15.4 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Smoke-free Days (Biochemically Verified) During a 7-day Quit Attempt.
Description: Day 17 will be the beginning of a 7-day quit attempt, during which the total number of days of abstinence will be assessed.
Time Frame: Days 17-23
Population: Number of subjects who completed the study in each arm
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 28 | 33
days | 3.6 (2.3) | 3.7 (2.3)

2. Secondary Outcome: Cognitive Performance
Description: Participants will complete neurocognitive tests designed to test working memory and attention. These tests are similar to computer games, in that participants will push a button in response to the pictures they see.
Time Frame: Baseline (Day 0), Day 14 (day before start of 24-hour abstinence period), Day 16 (after 24-hour abstinence period ends)
Population: Number of subjects who completed the study in each arm
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 28 | 33
number of correct responses
  Working memory (Baseline) | 47.3 (5.0) | 46.6 (5.6)
  Working memory (Day 14) | 49.0 (4.6) | 48.4 (5.1)
  Working memory (Day 16) | 49.3 (7.0) | 47.1 (6.9)
  Attention (Baseline) | 111.3 (8.9) | 103.4 (20.4)
  Attention (Day 14) | 113.9 (8.3) | 110.5 (11.3)
  Attention (Day 16) | 115.2 (6.4) | 111.0 (11.6)

3. Secondary Outcome: Subjective Symptoms
Description: Smoking urges [Questionnaire of Smoking Urges-Brief; QSU-B; 10-items rated on a 7-point scale (1=strongly disagree, 7=strongly agree) and summed for total score (range: 10-70). Higher scores=greater urge to smoke.] Negative mood [Negative Affect scale (10 items) from the Positive and Negative Affect Schedule; PANAS; 20-item Likert-format measure; The subscale was summed to create a summary score (range: 10-50); Lower negative affect indicates better outcomes.] Nicotine withdrawal [Minnesota Nicotine Withdrawal Scale-Revised; MNWS-R; 15 symptoms are rated on intensity with the following scale: 0=none, 1=slight, 2=mild, 3=moderate, 4=severe. The first 9 items are summed for total score (range: 0-36); higher scores=more severe withdrawal.].
  Measures assessed at the following visits: Baseline; Day 7 (monitoring visit); Day 14 (Day before 24-hour abstinence period), Day 16 (after 24-hour abstinence period), and Days 17-23 (7-day quit attempt).
Time Frame: Baseline (day 0), Days 7, 14, 16, 17, 19, 21, and 23
Population: Number of subjects who completed the study in each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 28 | 33
units on a scale
  Smoking urges (baseline) | 29.4 (13) | 30.2 (14.4)
  Smoking urges (day 7) | 21.6 (9.8) | 25.9 (15.4)
  Smoking urges (day 14) | 21.1 (13.2) | 24.1 (12.5)
  Smoking urges (day 16) | 33 (15.6) | 36 (17.3)
  Smoking urges (day 17) | 21.7 (9.9) | 29.7 (17.8)
  Smoking urges (day 19) | 20.7 (11.8) | 25.2 (14.1)
  Smoking urges (day 21) | 19.8 (9.6) | 22.2 (12.5)
  Smoking urges (day 23) | 18.8 (8.6) | 23.2 (14.2)
  Negative Mood (baseline) | 12.2 (2.9) | 12.7 (4.5)
  Negative Mood (day 7) | 11.2 (2.6) | 12.0 (3.7)
  Negative Mood (day 14) | 11.8 (3.5) | 11.9 (3.6)
  Negative Mood (day 16) | 13.7 (5.7) | 13.9 (4.4)
  Negative Mood (day 17) | 11.6 (3.5) | 11.7 (2.6)
  Negative Mood (day 19) | 11.6 (2.9) | 12.0 (2.9)
  Negative Mood (day 21) | 12.0 (3.6) | 11.8 (2.3)
  Negative Mood (day 23) | 11.1 (2.5) | 12.0 (3.6)
  Withdrawal (baseline) | 5 (2.8) | 5.6 (4.2)
  Withdrawal (day 7) | 4.6 (2.3) | 5.4 (4.5)
  Withdrawal (day 14) | 5.1 (3.8) | 3.9 (4.2)
  Withdrawal (day 16) | 7.6 (6.2) | 7.7 (5.7)
  Withdrawal (day 17) | 4.6 (4.4) | 4.6 (4.7)
  Withdrawal (day 19) | 5.2 (4) | 4.6 (4.5)
  Withdrawal (day 21) | 4.7 (3.5) | 4.8 (3.9)
  Withdrawal (day 23) | 3.2 (3.5) | 4.1 (5.0)

4. Secondary Outcome: Common Side Effects of Galantamine Check List
Description: Subjects completed a side effect checklist at every in-person study visit over the course of the treatment period. Subjects rated the severity of 37 common side effects of galantamine on the following scale: 0=none, 1=mild, 2=moderate, 3=severe. The average of all items was used to create a summary side effect score (range for total summary score 0-3). Higher scores indicate greater severity of side effects.
  Side effects of galantamine were assessed at the following in-person sessions: Baseline session; Day 7 (brief monitoring visit); Day 14 (Day before 24-hour abstinence period), Day 16 (after 24-hour abstinence period), and Days 17-23 (during the 7-day quit attempt).
Time Frame: Baseline (day 0), Days 7, 14, 16, 17, 19, 21, and 23
Population: Number of subjects who completed the study in each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Galantamine | Placebo
Number analyzed (Participants) | 28 | 33
units on a scale
  Baseline | .03 (.06) | .04 (.07)
  Day 7 | .09 (.09) | .07 (.08)
  Day 14 | .1 (.15) | .06 (.11)
  Day 16 | .1 (.12) | .08 (.1)
  Day 17 | .08 (.12) | .05 (.08)
  Day 19 | .07 (.09) | .05 (.09)
  Day 21 | .06 (.08) | .05 (.08)
  Day 23 | .05 (.06) | .05 (.08)

ADVERSE EVENTS:
Time Frame: 23 days
Arm/Group | Galantamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 4/40 | 3/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine (N=40) | Placebo (N=42)
Difficulty sleeping (General disorders) | 4 (10) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT01669538/Prot_SAP_000.pdf